CLINICAL TRIAL: NCT04741581
Title: Effect on Swallowing Function As Assessed by a Videofluoroscopy (VFS) One Day Study with Bolus of Various Viscosities, Followed, in a Subset of Patients, by an Acceptability 14 Days Study Combined with an Exploratory Hydration Assessment Study At a Prescribed Viscosity.
Brief Title: ThickenUp® Gel Express for Patients with Dysphagia
Acronym: HYDRA-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20.18.CLI
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-08

CONDITIONS: Dysphagia, Esophageal
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: prospective, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thicken up (Other): Assess the effect of ThickenUp® Gel Express at increasing viscosities (slightly thick, nectar, honey, and pudding) on swallowing function compared to water using VFS (N=100), in patients affected by Oropharyngeal dysphagia (OD).
  Interventions: Dietary Supplement: ThickenUp® Gel Express

INTERVENTIONS:
Dietary Supplement: ThickenUp® Gel Express — Thickening gel

SUMMARY:
Evaluation of swallowing function and hydration following consumption of ThickenUp® Gel Express in patients with dysphagia.

DETAILED DESCRIPTION:
ThickenUp® Gel Express for Patients With Dysphagia ("Hydra-01 Study"): Effect on Swallowing Function as Assessed by a Videofluoroscopy (VFS) One Day Study With Bolus of Various Viscosities (Study Part 1) and Followed, in a Subset of Patients, by a United Kingdom Advisory Committee on Borderline Substances (UK ACBS) Acceptability 14 Days Study Combined With an Exploratory Hydration Assessment Study at a Prescribed Viscosity (Study Part 2).

ELIGIBILITY:
Key inclusion criteria (for study part 1 and part 2):

1. Aged ≥ 18 years;
2. Diagnosed with oropharyngeal dysphagia and with a documented impaired safety of swallow by V-VST and PAS >1 during VFS;
3. History and/or current of swallowing difficulties;
4. Willing to adhere to the restrictions specified in the protocol;
5. Must be competent to understand the nature of the study and capable of giving written informed consent. In case patients are not capable of providing written informed consent (i.e. affected by dementia) a family/legal representative could provide the consent for the study.
6. Willing to report for the scheduled study visits and communicate to study personnel about adverse events and concomitant medication use.

Key exclusion criteria (for study part 1 and part 2):

1. Patients suffering from idiosyncratic phenomena or who are allergic to iodinated contrast media;
2. Major respiratory disease requiring oxygen or undergoing any type of surgery in the three months prior to the study;
3. Current diarrhea, vomiting or abdominal pain;
4. Alcohol or drug dependence (based on anamnesis only);
5. COVID-19 positive patients (with or without symptoms) at the time of enrolment;
6. Patients who, in the judgment of the investigator, are likely to be noncompliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
7. Having participated in a clinical study in the last 4 weeks and received compensation beyond a certain approved and predefined limit;
8. Having a clinical condition that is contraindicated with the study product;
9. Positive urine pregnancy test at screening for women of childbearing potential;
10. Allergy towards milk, mustard, egg, or celery.

Additional inclusion criteria for study part 2 only:

1. Patient willing to participate in study part 2;
2. Patient/caregiver able to record daily GI symptoms, compliance and fluid intake;
3. Patient able to respond to acceptability questionnaire (organoleptic properties, texture, appearance).
4. Patient willing to only use study product as the sole thickening agent during the Part 2.

Additional exclusion criteria for study part 2 only:

1. Undergone a major gastrointestinal surgery less than 3 months prior to enrolment in this study;
2. Obstruction of the gastrointestinal tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Score (PAS) | 1 day
  Part 1 -Bolus penetration into the laryngeal vestibule (PAS Score): the maximum PAS score across the different boluses assessed during videofluoroscopic (VFS) recording.
The United Kingdom Advisory Committee on Borderline Substances (UK ACBS) | 14 days
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Spain

IPD SHARING:
Plan to Share IPD: No